CLINICAL TRIAL: NCT03515928
Title: An Investigation of the Effects of Ultrasonic Noise Exposure on the Human Auditory System Via Pure Tone Audiometry (PTA) on Audiometrically Healthy Volunteers.
Brief Title: The Effects of Ultrasonic Noise Exposure on Human Hearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ultrahaptics Ltd (Industry)
Collaborators: Avon Partnership NHS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UH-PAN-001
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Hearing Loss
Keywords: Ultrasound, Hearing
MeSH Terms: conditions — Hearing Loss | interventions — Audiometry, Pure-Tone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noise Exposed Group (Active Comparator)
  Interventions: Other: Ultrasonic noise exposure; Diagnostic Test: Pure Tone Audiometry
- Control Group (Placebo Comparator)
  Interventions: Diagnostic Test: Pure Tone Audiometry

INTERVENTIONS:
Other: Ultrasonic noise exposure — Group will be exposed to 40kHz ultrasonic noise at 110-120 dB SPL for 15 minutes.
  Arms: Noise Exposed Group
Diagnostic Test: Pure Tone Audiometry — Participants will undergo 2 (pre and post exposure) hearing tests

SUMMARY:
The aim of this research is to investigate the effects of ultrasonic noise exposure on the human auditory system (how it effects hearing). Current international regulations concerning ultrasound exposure differs significantly and are based on scarce and outdated scientific data; hence the motivation for this research. A cohort of 20 audiometrically healthy volunteers will undergo pure tone audiometry (PTA); a standard test for hearing sensitivity, at both pre and post exposure to ultrasonic noise (40kHz for 15 min at 120 dB SPL). A subgroup of 10 subjects will be used as a control group. The resulting audiograms will establish the extent of any recoverable loss in hearing sensitivity known as temporary threshold shifts (TTS).

ELIGIBILITY:
Inclusion Criteria:

* Adult, audiometrically healthy

Exclusion Criteria:

* Underlying/pre-existing hearing impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Temporary Threshold Shifts (TTS) | Audiometry will be conducted immediately (with 2 hours) from noise exposure
  Mild and recoverable hearing loss in sensitivity due to noise exposure will be checked for statistical significance using paired and independent t-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrahaptics, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided